CLINICAL TRIAL: NCT05848843
Title: A Phase I Study of Adagrasib and Durvalumab for Treatment of Advanced Non-small Cell Lung Cancers and Gastro-intestinal Cancers Harboring KRAS G12C Mutations
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: 0 participant accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: AstraZeneca (Industry); Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0782; NCI-2023-03640 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-04-28; First posted 2023-05-08 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer; Gastro-intestinal Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — durvalumab; adagrasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Confirmation Cohort (Experimental)
  Interventions: Drug: Durvalumab; Drug: Adagrasib
- Dose Expansion Cohort (Experimental)
  Interventions: Drug: Durvalumab; Drug: Adagrasib

INTERVENTIONS:
Drug: Durvalumab — Given by vein (IV)
Drug: Adagrasib — Given by PO

SUMMARY:
To find a recommended dose of the combination of adagrasib and durvalumab that can be given to patients with cancers that have a KRAS G12C mutation.

DETAILED DESCRIPTION:
Primary Objectives:

• To determine the safety and tolerability, and to establish the recommended dose of the adagrasib and durvalumab combination in advanced NSCLC or GI cancer patients.

Secondary Objectives:

* To determine the objective response rate of the adagrasib and durvalumab combination for frontline treatment of advanced NSCLC harboring a KRAS G12C mutation.
* To determine the objective response rate of the adagrasib and durvalumab combination for treatment of advanced CRC that have progressed on prior therapy with KRAS G12C inhibitors.
* To determine duration of response (DOR) and progression-free survival (PFS) for the combination of the adagrasib and durvalumab in patients with advanced NSCLC harboring a KRAS G12C mutation.
* To determine DOR and PFS for the combination of the adagrasib and durvalumab in patients with advanced CRC that have progressed on prior therapy with KRAS G12C inhibitors.

Exploratory Objectives:

* To assess predictive biomarkers of response and resistance to the combination of adagrasib and durvalumab.
* To assess mechanisms of tumor cell adaptation upon treatment with the combination of adagrasib and durvalumab.
* To determine mechanisms of acquired resistance to the combination of adagrasib and durvalumab.
* To assess the effect of the combination of adagrasib and durvalumab on the immune tumor microenvironment.
* To generate cell lines and patient derived xenograft (PDX) models from tumor samples.
* To assess the anti-tumor reactivity of tumor infiltrating lymphocytes (TIL) from tumor biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. For the dose confirmation cohort, histologically confirmed diagnosis of NSCLC or carcinomas of gastro-intestinal tract, including, but not limited to, colorectal adenocarcinoma, pancreatic adenocarcinoma, and cholangiocarcinoma. For the Dose Expansion cohorts, only NSCLC and colorectal adenocarcinoma histologies are eligible.
2. Presence of KRAS G12C mutation detected by assay performed in a CLIA-certified environment.
3. Metastatic disease or locally advanced disease not amenable to local therapy.
4. ECOG performance status 0 or 1.
5. Presence of measurable disease per RECIST v1.1.
6. Any number of prior lines of therapy, including prior KRAS G12C inhibitor. For the Dose Expansion cohorts, only treatment naïve NSCLC patients and colorectal adenocarcinoma patients with disease progression on prior KRAS G12Ci are eligible. NSCLC patients that completed curative intent treatment of their disease ≥6 months prior to enrollment are eligible for frontline expansion cohort as long as they have not been previously treated with a KRAS G12C inhibitor.
7. Age ≥ 18 years.
8. Life expectancy of at least 3 months.
9. Most recent prior systemic therapy (e.g., chemotherapy, immunotherapy or, investigational agent) and radiation therapy discontinued at least 2 weeks before first dose date.
10. Recovery from the adverse effects of prior therapy at the time of enrollment to ≤ Grade 1 (excluding alopecia and parameters superseded by other eligibility criteria [eg, laboratory parameters]).
11. Laboratory values within the screening period:

    * Absolute neutrophil count ≥ 1,000/mm3 (≥ 1.0 x 109/L)
    * Platelet count ≥ 100,000/mm3 (≥ 100 x 109/L)
    * Hemoglobin ≥ 9 g/dL
    * Total bilirubin ≤ 1.5 x Upper Limit of Normal (ULN) (if associated with liver metastases or Gilbert's disease, ≤ 3 x ULN)
    * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 x ULN (if associated with liver metastases, ≤ 5 x ULN)
    * Creatinine clearance ≥50 mL/min calculated using a validated prediction equation (e.g., Cockcroft-Gault, MDRD, or 24-hour urine CrCl).
12. Women of child-bearing potential (WOCBP) or men whose partner is a WOCBP agrees to use contraception while participating in this study, and for a period of 6 months following termination of study treatment (see Reproductive Health below).
13. Completed informed consent process, including signing IRB/EC-approved informed consent form.
14. Willing to comply with clinical trial instructions and requirements. Reproductive Health

Patients who are biologically capable of having children and sexually active must agree to use an acceptable method of contraception for the duration of the treatment period and for at least 6 months after the last dose of study treatment. The Investigator will counsel the patient on selection of contraception method and instruct the patient in its consistent and correct use. Examples of acceptable forms of contraception include:

* Oral, inserted, injected or implanted hormonal methods of contraception, provided it has been used for an adequate period of time to ensure effectiveness.
* Correctly placed copper containing intrauterine device (IUD).
* Male condom or female condom used WITH a spermicide.
* Male sterilization with confirmed absence of sperm in the post-vasectomy ejaculate.
* Bilateral tubal ligation or bilateral salpingectomy. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control.

The Investigator will instruct the patient to call immediately if the selected birth control method is discontinued or if pregnancy is known or suspected.

Note: Women are considered post-menopausal and/or not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical

Exclusion criteria:

1. Radiation to the lung >30 Gy within 3 months prior to the first dose of study treatment.
2. Active brain metastases. Patients are eligible if brain metastases are adequately treated and patients are neurologically stable for at least 2 weeks prior to the first dose of study treatment without the use of corticosteroids or are on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent).
3. Carcinomatous meningitis.
4. History of significant hemoptysis or hemorrhage within 4 weeks of the first dose date.
5. Active or prior documented autoimmune or inflammatory disease, as follows:

   * Inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
   * History of interstitial lung disease (ILD) or radiation pneumonitis requiring steroid treatment, or any evidence of clinically active ILD or pneumonitis.
   * Other medically important autoimmune disease within 2 years prior to the first dose of study treatment. NOTE: Patients with Type 1 diabetes, vitiligo, Graves' disease requiring only hormone replacement, hypothyroidism, or psoriasis not requiring systemic treatment within the past 2 years are not excluded.
6. Immunocompromising conditions, as follows:

   * Use of immunosuppressive medication within 28 days prior to the first dose of study treatment, with the exceptions of corticosteroids.
   * History of primary immunodeficiency.
   * History of allogeneic transplant.
7. Receipt of a live vaccine within 30 days prior to first dose of study treatment.
8. Known severe hypersensitivity to study drugs and/or any of its excipients.
9. Known human immunodeficiency virus (HIV) infection or acute or chronic hepatitis B or C infection. Patients treated for hepatitis C with no detectable viral load are permitted.
10. Major surgery within 4 weeks prior to first dose of study treatment.
11. History of intestinal disease or major gastric surgery likely to alter absorption of study treatment or inability to swallow oral medications.
12. Any of the following cardiac abnormalities:

    * Unstable angina pectoris or myocardial infarction within the past 6 months.
    * Symptomatic or uncontrolled atrial fibrillation within the past 6 months.
    * Congestive heart failure ≥NYHA Class 3 within the past 6 months.
    * Prolonged QTc interval >480 milliseconds, or immediate family or medical history of congenital Long QT Syndrome.
13. History of stroke or transient ischemic attack within 6 months prior to first dose of study treatment.
14. Ongoing need for a medication with any of the following characteristics that cannot be switched to alternative treatment prior to study entry: known risk of QT prolongation or Torsades de Pointes; substrate of CYP3A with narrow therapeutic index; strong inducer of CYP3A and/or P-gp; strong inhibitor of BCRP; and proton pump inhibitors (see Appendix 2).
15. Known or suspected presence of another malignancy that could be mistaken for the malignancy under study during disease assessments.
16. Pregnancy. WOCBP must have a negative serum or urine pregnancy test documented within the screening period prior start of study drug.
17. Breast-feeding or planning to breast feed during the study or within 6 months after the last dose of study treatment.
18. Any serious illness, uncontrolled inter-current illness, psychiatric illness, active or uncontrolled infection, or other medical history, including laboratory results, which, in the Investigator's opinion, would be likely to interfere with the patient's participation in the study, or with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo V. Negrao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org